CLINICAL TRIAL: NCT02195258
Title: Pharmacogenetic of the Salbutamol Efficacy in Asthma Crisis for Children in Emergency Department
Brief Title: Pharmacogenetic of Salbutamol in Pediatric Asthma Crisis
Acronym: Pegase
Status: Completed | Type: Observational
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Helene Chappuy, MD Ph D, Hôpital Necker-Enfants Malades
Other Study IDs: URC Paris centre
Record Dates: First submitted 2013-07-04; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Saliva from patient were collected using Oragen®.DNA OG-500 kit, (DNA Genotek, Kanata, Canada) or swabs (Catch-All™ sample collection swabs from Epicentre Biotechnologies, Madison, WI), and stored at room temperature or -20°C, respectively.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- salbutamol

SUMMARY:
this study is designed to identify the genetic factors which can be implicated in the salbutamol responsiveness for asthmatic children in pediatric emergency department

DETAILED DESCRIPTION:
Patients from 6 to 16 years old consulting for an acute asthma exacerbation and receiving a treatment by salbutamol according to the usual care could be recruited.Saliva from patient were collected using Oragen®.DNA OG-500 kit or swabs.Based on literature review, four SNP were chosen:ADBR2 gene), ARG gene, and GSNOR gene.

ELIGIBILITY:
Inclusion Criteria:

* children
* 6-16 years old
* asthmatic patients
* consulting for an exacerbation in a pediatric emergency department
* parental informed consent

Exclusion Criteria:

* comorbidity
* peak flow no available
* pneumonia

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 6-16 years old asthmatic patients consulting for an exacerbation in a pediatric emergency department
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
pre- and post-bronchodilator FEV1 value (BDR = 100 x [post-FEV1 - pre-FEV1]/pre-FEV1) | Day 0
  comparison of acute response to salbutamol calculated as the percentage difference between the pre- and post-bronchodilator FEV1 value (BDR = 100 x [post-FEV1 - pre-FEV1]/pre-FEV1) between the different polymorphism

SECONDARY OUTCOMES:
polymorphism on the response delay | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Chappuy, MDPhD, Principal Investigator — APHP
Locations (1):
- Necker Enfants Malades Hospital, Paris, France